CLINICAL TRIAL: NCT06327919
Title: Effects of Probiotic Supplementation With Weight Reducing Plan on Anthropometric Measures, Body Composition, Eating Behavior, and Related Hormone Levels in Patients With Food Addiction and Weight Regain After Bariatric Surgery: A Randomized Clinical Trial
Brief Title: Effects of Probiotic Supplementation With Weight Reducing Plan in Patients With Food Addiction and Weight Regain After Bariatric Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Nutrition and Food Technology Institute (Other)
Responsible Party: Principal Investigator, Dr Azita Hekmatdoost, Principal Investigator, National Nutrition and Food Technology Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 62885
Record Dates: First submitted 2024-03-18; First posted 2024-03-25 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Weight Regain After Bariatric Surgery and Food Addiction
MeSH Terms: conditions — Food Addiction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Probiotic supplementation with a weight loss program and ten one-hour online individual sessions cognitive behavioral therapy for 12 weeks.
  multi-strain probiotics were used in this study. Each probiotic capsule contains Lactobacillus acidophilus, Bifidobacterium bifidum, Bifidobacterium lactis, Bifidobacterium longum, Lactobacillus reuteri, Lactobacillus rhamnosus, magnesium stearate and maltodextrin. 1.8 × 109 CFU / capsule. 2 capsules per day, for 12 weeks.
  Interventions: Dietary Supplement: Probiotic supplement
- Placebo (Placebo Comparator): Placebo supplementation with a weight loss program and ten one-hour online individual sessions cognitive behavioral therapy for 12 weeks.
  The placebo capsule contains 300 mg of starch. 2 capsules per day, for 12 weeks
  Interventions: Other: Placebo supplement

INTERVENTIONS:
Dietary Supplement: Probiotic supplement — multi-strain probiotics were used in this study. Each probiotic capsule contains Lactobacillus acidophilus, Bifidobacterium bifidum, Bifidobacterium lactis, Bifidobacterium longum, Lactobacillus reuteri, Lactobacillus rhamnosus, magnesium stearate and maltodextrin. 1.8 × 109 CFU / capsule. 2 capsules per day, for 12 weeks
  Arms: Intervention
Other: Placebo supplement — The placebo capsule contains 300 mg of starch. 2 capsules per day, for 12 weeks
  Arms: Placebo

SUMMARY:
To study the effects of probiotic supplementation with a weight loss program and cognitive behavioral therapy (CBT) on anthropometric measures, eating behavior, food addiction, and related hormone levels in patients with food addiction and weight regain after bariatric surgery, 50 patients who referred to obesity clinic with weight regain (regaining ≥10% nadir weight) after bariatric surgery (at least 18 months), and food addiction will be randomly allocated to receive a weight loss program and CBT plus either probiotic, or placebo for 12 weeks. At the first and the end of the intervention, anthropometric measurements, eating behavior, food addiction, leptin, serotonin, and oxytocin will be assessed and compared between groups.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥25 kg/m2; willingness to participate in the study; not having diseases such as cancer, thyroid, diabetes, renal or liver (except fatty liver); non-pregnant or lactating or menopause or professional athlete; not use of any antibiotics in the last three weeks and any protein or probiotic supplement in the last month

Exclusion Criteria:

* taking antibiotic; using probiotic supplements/products or protein supplements; using weight-loss or appetite-suppressing medications; pregnancy; consuming less than 90% of the supplements prescribed during the study; following less than 90% of diet or physical activity for more than 10 days; participants who refuse to continue the study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-05-25 (Actual); Study Completion 2023-09-23 (Actual)

PRIMARY OUTCOMES:
Weight | 12 weeks
  According to changes in body weight
BMI | 12 weeks
  According to changes in BMI
Waist circumference | 12 weeks
  According to changes in waist circumference
Fat mass | 12 weeks
  According to changes in body fat mass
Food addiction | 12 weeks
  According to changes in Score Of Yale Food Addiction Scale questionnaire

SECONDARY OUTCOMES:
Eating behavior | 12 weeks
  According to changes in Score Of Three-Factor Eating Questionnaire
Leptin | 12 weeks
  According to changes in serum level of leptin
Serotonin | 12 weeks
  According to changes in serum level of serotonin
Oxytocin | 12 weeks
  According to changes in serum level of oxytocin

CONTACTS AND LOCATIONS:
Locations (2):
- Iran (2):
  - Azita Hekmatdoost, Tehran, Middle East
  - National Nutrition and Food Technology Research Institute, Tehran

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification will be shared.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: beginning 9 months and ending 36 months following article publication.
Access Criteria: send mail to Atoosa.saidpour@gmail.com.